CLINICAL TRIAL: NCT06628297
Title: Small Vessel Disease of the Brain and Heart a PET Perfusion Study of Training Effects
Brief Title: Comparison of Differencens in VO2-max, Perfusion of the Heart and Brain and Cognitive Performance Between Patients with Type 2 Diabetes and Healthy Age Matched Controls.
Acronym: SVAT
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Collaborators: Danish Cardiovascular Academy (Unknown); Bispebjerg Hospital (Other); The Dagmar Marshall Foundation (Other); Steno Diabetes Center Copenhagen (Other)
Responsible Party: Principal Investigator, Thomas Ehlig Hjermind Justesen, Principal Investigator, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: PhD2024013-HF; PhD2024013-HF (Other Grant/Funding Number: Danish Cardiovascular Academy)
Record Dates: First submitted 2024-09-30; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Microvascular Disease; Microvascular Complications; Dementia; Diabetes Mellitus Type 2; Cerebral Hypoperfusion
Keywords: microvascular disease; microvascular complications of the heart; microvascular complications of the brain; diabetes type 2; dementia; microvascular disease patophysiology
MeSH Terms: conditions — Dementia; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — We will keep bllod samples in a Biobank. Currently, the relevant tests are not available yet. But once they are, we will use the blood samples to look at markers of neurological damage and inflammation and are associated with dementia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 48 patients with type 2 diabetes and increased risk of microvascular disease: Baseline measurements of:
  * [15O]H2O PET of heart and brain
  * Blood sampling
  * Echocardiography
  * Brain MRI
  * Cognitive tests
  * Cardiorespiratory fitness test
  * Muscular function test
  Interventions: Diagnostic Test: PET
- 24 healthy age-matched participants: Baseline measurements of:
  * [15O]H2O PET of heart and brain
  * Blood sampling
  * Echocardiography
  * Brain MRI
  * Cognitive tests
  * Cardiorespiratory fitness test
  * Muscular function test
  Interventions: Diagnostic Test: PET

INTERVENTIONS:
Diagnostic Test: PET — PET imaging will be performed with a Discovery 710 PET/CT scanner (GE Healthcare, Milwaukee, WI, USA). Four 5-minute PET recordings will be performed of each subject within a single scanning session of 70 min. Two consecutive 5-minute scans are conducted of the heart and brain in rest. [15O]H2O, is produced on-site (GENtrace, GE, Uppsala, Sweden), and 600 MBq [15O]H2O is intravenously injected by an automatic Hidex Radiowater Generator (Hidex, Turku, Finland). To induce heart vasodilation, adenosine is infused (140 g/kg/min) for 6 min and a scan of the heart is repeated. To induce brain vasodilation, 1 g of acetazolamide is infused over 5 min and 15 min later the brain is scanned. Myocardial perfusion is calculated using CarimasCE software version 1.3.1. (Turku, Finland). Cerebral perfusion is calculated using PMOD software (PMOD Technologies, Switzerland).
  Other Names: MRI; VO2-max; cognitive testing

SUMMARY:
In the aging population, ischemic heart disease, stroke and dementia are increasingly prevalent. Diagnosis and treatment of the former two i.e., large-vessel coronary heart disease and endovascular thrombectomy of the brain in relation to stroke have improved significantly. Yet, the majority of elderly patients with ischemic heart disease do not have large-vessel heart disease and it seems that small vessel disease (SVD) may explain a large fraction of these cases as well as the cardiovascular morbidity in the elderly. Hence, the current development in diagnostics and treatments of ischemic heart disease does not address the most common subtype of ischemic disease seen in elderly patients.

It has been suggested that SVD is part of a multisystem disorder and several systematic reviews have addressed the hypothesis of a potential link between small vessel disease of the heart, brain, and kidneys. Cerebral SVD is prevalent in the aging population causing cognitive impairment, dementia, and an increased risk of stroke, and cerebral hypoperfusion is an acknowledged cause of vascular dementia and a possible cause of Alzheimer's disease. Further, cognitive impairment within multiple cognitive domains is highly prevalent in heart failure and is associated to an increased risk of dementia. The link between heart failure and dementia may be due to multisystem SVD, although a direct link between the two is possible.

Among other known risk factors such as age, hypertension, and female sex, diabetes is a major cause of SVD and is linked to coronary heart disease as well as cognitive impairment. The diagnosis of cerebral SVD relies on MRI detecting infarctions, haemorrhages, microbleeds and ischemic white matter changes, i.e. Fazekas score. In contrast, perfusion PET is used to image myocardial perfusion in patients with coronary SVD; and coronary SVD is recognized as a part of the pathophysiology in angina, coronary artery disease, and heart failure. Perfusion PET before and after adenosine-induced vasodilation allows for measuring, the myocardial flow reserve (MFR), i.e. perfusion capacity, which in the absence of regional perfusion defects, is a measure of coronary SVD. Prof. Eva Prescott have recently shown that reduced MFR obtained by 82Rb PET is a strong predictor of future microvascular events and all-cause mortality.

Exercise is well known to improve cognitive health but professor Carl-Johan Boraxbekk has shown that the effect on cognitive performance may be dependent on the initial cerebrovascular status, as patients with moderate to severe white matter changes did not improve after a 6 months physical activation intervention in contrast to patients with mild changes. Yet, it is possible to improve brain function in diabetic patients through either dietary or exercise interventions.

Systemic SVD is measured as cerebral SVD (reduced brain perfusion during acetazolamide-induced vasodilation) and coronary SVD (reduced heart perfusion during adenosine-induced vasodilation). The researchers anticipate that patients with type 2 dabetes have reduced perfusion capacity of the brain and heart correlating to reduced cognition and cardiorespiratory fitness (VO2-max).

DETAILED DESCRIPTION:
The goal of this clinical trial is to compare baseline measurements relevant to microvascular disease between patients with diabetes and increased risk of microvascular disease with healthy age-matched control.

The researchers wish to examine if small vessel disease is a disease that affects several organs at once in the same individuals by examining it in the brain and heart in the same participants. The researchers will also test if cardiorespiratory conditioning (VO2-max), blood perfusion to the heart and brain and cognitive performance are correlated in patients with microvascular disease.

To adress these aims the researchers have defined the following assumptions that they will refute or confirm through this study:

* Patients with type 2 diabetes and increased risk of small vessel disease have significantly reduced perfusion capacity of the brain and heart compared to healthy controls as part of a multisystem disease
* Perfusion capacity of the brain and heart, the cardiorespiratory fitness level of the subjects and cognitive performance are directly linked.

  48 patients with diabetes and 24 healthy age-matched controls will undergo baseline testing that include:
* Cardiopulmonal Exercise Test (CPET) to determine cardiopulmonal conditioning (VO2-max)
* Isometric knee strength (if logistically possible)
* Echocardiography
* Blood perfusion capacity of the heart and brain via [15O]H2O-PET scans
* Brain MRI to determine structural damages
* Blood samples for basic health check (relevant to inclusion, exclusion and safety) and blood samples looking at endothelial and neurological damage for a biobank
* Cognitive testing (SCIP-D and CANTAB)

Afterwards the researchers will compare the results between the two groups and see if there is a correlation between VO2-max, blood perfusion to the heart and brain and cognitive performance.

ELIGIBILITY:
Inclusion Criteria for the patients with type 2 diabetes:

Diabetes type II diagnose with one of the following:

* Duration over 5 years
* Moderate microalbuminuria
* Non-proliferative diabetic retinopathy

  * Speaks and understands Danish (required for reliable cognitive testing)
  * Able to provide informed and written consent

Exclusion Criteria or the patients with type 2 diabetes:

Moderate to high intensity training >1 times/week.

* Previous AMI, atrial fibrillation, significant cardiac valve disease, HFrEF (LVEF <45%), asthma.
* Previous stroke or significant neurological disease including cognitive dysfunction.
* Ongoing depression.
* Hypothyroidism
* Unable or unwilling to participate in training, e.g., due to injury, arthrosis or lung disease.

Inclusion Criteria for the healthy age-matched controls:

* Age > 60 years
* No diagnosis of T2D according to WHO's criteria.
* Speaks and understands Danish (required for reliable cognitive testing)
* Able to provide informed and written consent

Exclusion Criteria for the healthy age-matched controls:

* Moderate to high intensity training >2 times/week.
* Previous AMI, atrial fibrillation, significant cardiac valve disease, HFrEF (LVEF <45%), asthma.
* Previous stroke or significant neurological disease including cognitive dysfunction.
* Ongoing depression.
* Hypothyroidism
* Unable or unwilling to participate in training, e.g., due to injury, arthrosis or lung disease.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes with increased risk of microvascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
[15O]H2O PET assessment of the blood perfusion to the brain | From baseline testing to end of study, 6 months
  We will use the scan to determine our primary outcome: Blood perfusion to the brain. Radioactive water ([15O]H2O) will be used as a PET-tracer since it follows the blood and is the gold standard tracer for PET-based blood perfusion measurements. We measure the blood perfusion of both the brain as the perfusion capacity, meaning the difference between blood perfusion to the organ at rest and the maximally possible perfusion. In the brain we use injection of diamox to stimualte maximal dilation of the cerebral arteries which corresponds to the maximally possible perfusion of the brain.
[15O]H2O PET assessment of the blood perfusion of the heart | From baseline testing to end of study, 6 months
  We will use the scan to determine our primary outcome: Blood perfusion to the heart.
  Radioactive water ([15O]H2O) will be used as a PET-tracer since it follows the blood and is the gold standard tracer for PET-based blood perfusion measurements.
  We measure the blood perfusion of both the heart as the perfusion capacity, meaning the difference between blood perfusion to the organ at rest and the maximally possible perfusion. In the heart we use injection of adenosin to stimualte maximal dilation of the coronary arteries which corresponds to the maximally possible perfusion of the heart.

SECONDARY OUTCOMES:
Cognitive performance (CANTAB) | From baseline testing to end of study, 6 months
  Testing of a broad range of cognitive functions. The test is tablet based and one of the most "investigator-independent" cognitive tests available. The test takes around 45 minutes to perform.
Cognitive Performance (SCIP-D) | From baseline testing to end of study, 6 months
  Assessed via SCIP-D in order to evaluate a broad range of cognitive areas in around 15-20 minutes. Both groups will undergo both tests. The primary investigator will receive learning in how to carry out the SCIP-D correctly.
  SCIP-D is a more clinically relevant test that can be used in a clinical setting to identify patients with cognitive dysfunction.
Cardiorespiratory fitness (VO2-max) | From baseline testing to end of study, 6 months
  Will be assessed as the maximal or peak oxygen consumption (VO2-max or VO2-peak) during a cardiopulmonal exercise test (CPET).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas EHJ Primary Investigator, Medical Doctor, Principal Investigator — University Hospital Bispebjerg and Frederiksberg
Locations (1):
- Bispebjerg and Frederiksberg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Have not gotten the necessary clearence